CLINICAL TRIAL: NCT03181841
Title: Effects of PF-06412562 on Value-based Decision-making in Healthy Individuals: a Mono-center, Randomized, Placebo Controlled, Double-blind Study (Phase I)
Brief Title: Effects of PF-06412562 on Value-based Decision-making in Healthy Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PHA-16-D1AGO-01
Record Dates: First submitted 2017-05-12; First posted 2017-06-09 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Decision Making

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active dose 1 (Experimental): Single dose of PF-06412562 in low dosage strength
  Interventions: Drug: PF-06412562
- Active dose 2 (Experimental): Single dose of PF-06412562 in medium dosage strength
  Interventions: Drug: PF-06412562
- Active dose 3 (Experimental): Single dose of PF-06412562 in higher dosage strength
  Interventions: Drug: PF-06412562
- Placebo (Placebo Comparator): Single dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06412562 — double-blind oral intake of single doses of the aforementioned drug or placebo
  Arms: Active dose 1; Active dose 2; Active dose 3
Drug: Placebo — double-blind oral intake of single doses of the aforementioned drug or placebo
  Arms: Placebo

SUMMARY:
Numerous psychiatric and neurodegenerative diseases like schizophrenia, dependency on drugs of abuse, depression and Parkinson's disease are related to motivational and cognitive deficits in value-based decision making, which frequently persist even after a successful pharmacological treatment. According to current neurobiologic models, cortical dopamine D1 receptors play a crucial role in taking value-based decisions. In this study, it will be investigated whether value-based decisions in healthy volunteers can be improved by stimulation of D1-receptors. For this purpose, a newly developed dopamine D1-agonist will be used, which selectively increases the activities of frontal D1- and D5-receptors. In this double-blind, randomized, placebo-controlled study, the effects of different single doses of PF-06412562, a not yet licensed D1-agonist, on value-based decision making will be compared with placebo. The use of different dosage strengths will allow to investigate a potential relationship between the extent of activity of the D1-receptor and its influence on behavioral indices.

Therefore, four parallel groups will be investigated. Each participant takes in a single dose of either PF-06412562 in different doses or placebo. A screening exam will be carried out 1-3 weeks before the drug intake, and a follow-up examination will be carried out approx. 1 week after the drug intake. At all 3 visits in the study centre, several tests for the investigation of value-based decision making will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature on the informed consent form
* Physically and psychiatrically healthy men and women
* Male and female subjects of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 28 days for females and 90 days for males after the last dose of assigned treatment. A subject is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children.
* Female subjects of non childbearing potential must meet at least one of the following criteria:

  * Have undergone a documented hysterectomy and/or bilateral oophorectomy;
  * Have medically confirmed ovarian failure or;
  * Achieved post menopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level confirming the post menopausal state.
* All other female subjects (including females with tubal ligations and females that do NOT have a documented hysterectomy, bilateral oophorectomy and/or ovarian failure) will be considered to be of childbearing potential.
* Aged 18-35 years
* Negative pregnancy test (see exclusion criteria)
* Normal or corrected-to-normal vision

Exclusion Criteria (selected):

* Pregnant female subjects; breastfeeding female subjects
* considered to be healthy based on an extensive pre-study screening including anamnesis, physical examination, laboratory investigations, vital signs, ECG, etc.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in a delay discounting task. | 1-3 weeks before (= baseline), 5 hours after, and approx. 1 week after drug intake.
  This validated computer-based decision-making test will be filled in by each participant at three time points during the study: 1-3 weeks before, 5 hours after, and approx. 1 week after a single oral intake of 1 out of 3 possible doses of PF-06412562, or matching placebo.
Change from baseline in a risk discounting task. | 1-3 weeks before (= baseline), 5 hours after, and approx. 1 week after drug intake.
  This validated computer-based decision-making test will be filled in by each participant at three time points during the study: 1-3 weeks before, 5 hours after, and approx. 1 week after a single oral intake of 1 out of 3 possible doses of PF-06412562, or matching placebo. It will be carried out after the test for outcome 1.
Effect of PF-06412562 on an effort discounting task (compared to placebo). | 5 hours after drug intake.
  This validated computer-based decision-making test will be completed by each participant 5 hours after a single oral intake of 1 out of 3 possible doses of PF-06412562, or matching placebo and after having completed the tests for outcome 1 and 2.
Effect of PF-06412562 on the Pavlovian to instrumental transfer task (compared to placebo). | 5 hours after drug intake.
  This validated computer-based decision-making task tests Pavlovian acquisition and transfer. It will be carried out by each participant immediately after the test in outcome 3.
Effect of PF-06412562 on an exploration / exploitation task (compared to placebo). | 5 hours after drug intake.
  This validated computer-based decision-making task tests different aspects of value-based decision making. It will be carried out by each participant immediately after the test in outcome 4.
Effect of PF-06412562 on a probabilistic reversal learning task (compared to placebo). | 5 hours after drug intake.
  This validated computer-based decision-making task tests different aspects of value-based decision making. It will be carried out by each participant immediately after the test in outcome 5.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability of PF-06412562) | throughout the study and up to 1 week after study drug intake.
  continuous assessment of adverse events by non-leading questions, repeated safety laboratory tests, repeated ECGs, repeated control of vital parameters.

OTHER OUTCOMES:
Plasma concentrations of PF-06412562 | blood sampling 4 hours and 8 hours after the study drug intake.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Tobler, Prof. Dr., Study Director — University of Zurich, Dept. of Economics; Alexander Jetter, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Dept. of Clinical Pharmacology and Toxicology, Zurich, Switzerland

REFERENCES:
- [Result] Soutschek A, Gvozdanovic G, Kozak R, Duvvuri S, de Martinis N, Harel B, Gray DL, Fehr E, Jetter A, Tobler PN. Dopaminergic D1 Receptor Stimulation Affects Effort and Risk Preferences. Biol Psychiatry. 2020 Apr 1;87(7):678-685. doi: 10.1016/j.biopsych.2019.09.002. Epub 2019 Sep 12. PMID 31668477
- [Result] Soutschek A, Kozak R, de Martinis N, Howe W, Burke CJ, Fehr E, Jetter A, Tobler PN. Activation of D1 receptors affects human reactivity and flexibility to valued cues. Neuropsychopharmacology. 2020 Apr;45(5):780-785. doi: 10.1038/s41386-020-0617-z. Epub 2020 Jan 21. PMID 31962344
- [Derived] Soutschek A, Tobler PN. A process model account of the role of dopamine in intertemporal choice. Elife. 2023 Mar 8;12:e83734. doi: 10.7554/eLife.83734. PMID 36884013